CLINICAL TRIAL: NCT07262320
Title: Epidemiology and Processes of Care for Renal Replacement Therapy in Acute Kidney Injury in Latin America
Acronym: LATAM-AKID
Status: Not yet recruiting | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Vantive Health LLC (Industry)
Responsible Party: Principal Investigator, Javier A. Neyra, Professor of Medicine, University of Alabama at Birmingham
Other Study IDs: IRB-300013633; IIR from Vantive (Other Grant/Funding Number: Vantive)
Record Dates: First submitted 2025-11-17; First posted 2025-12-03 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Dialysis; Critically Ill Acute Kidney Injury; Renal Replacement Therapy for Acute Kidney Injury in ICU; Acute Kidney Injury; Renal Replacement Therapy; AKI
Keywords: AKI; ICU; RRT; Latin America; acute kidney injury; renal replacement therapy; intensive care unit; dialysis
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute kidney injury patients requiring renal replacement therapy: Critically ill adult patients with acute kidney injury undergoing any form of renal replacement therapy in Latin American hospitals

SUMMARY:
This is an international, multicenter, observational study aimed at investigating acute kidney injury requiring renal replacement therapy (AKI-RRT) in Latin American countries. The main questions this study aims to answer are:

* What is the epidemiology, outcomes, and processes of care for patients with AKI-RRT in Latin America?
* How do outcomes differ across different countries in Latin America?
* What factors (demographics, clinical, socioeconomic) influence outcomes in patients with AKI-RRT in Latin America?

The main aims of this study are to:

* Establish a comprehensive database containing clinical, laboratory, treatment, process, and outcome data of patients with AKI-RRT in Latin America
* Describe current epidemiology of AKI-RRT in Latin America
* Compare processes of care and outcomes across different countries in Latin America
* Provide data resources to facilitate and promote clinical research in AKI-RRT

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (≥18) admitted to the ICU
* First ICU admission during current hospitalization
* Diagnosis of acute kidney injury stage 3 according to KDIGO guidelines
* RRT initiated no earlier than 3 days before or no later than 7 days after ICU admission

Exclusion Criteria:

* Transfer from outside hospital with ongoing RRT
* RRT exposure of less than 2 days (if CRRT or PD was provided) or less than 2 HD/SLED sessions
* Kidney failure (ESRD) patients on maintenance dialysis
* Kidney transplant recipients
* Previous or new diagnosis of glomerulonephritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients with AKI requiring RRT in Latin American countries
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
In-hospital mortality | From enrollment to hospital discharge or 90 days (whichever occurs first)
  The variable is coded as 1 = deceased and 0 = alive by the time of hospital discharge

SECONDARY OUTCOMES:
ICU mortality | From enrollment to ICU discharge or 90 days (whichever occurs first)
  The variable is coded as 1 = deceased and 0 = alive by the time of ICU discharge
90-day follow-up mortality | From enrollment to 90-days post-ICU admission follow-up
  The variable is coded as 1 = deceased and 0 = alive by the time of 90-day follow-up
Length of stay in the ICU | From ICU admission to death or ICU discharge (truncated at 90 days)
  Length of stay will be calculated as the total number of full days between admission and discharge from the ICU. A calendar day will be counted toward the total only if the duration of stay on that day is two hours or longer.
Length of stay in the hospital | From hospital admission to death or hospital discharge (truncated at 90 days)
  Length of stay will be calculated as the total number of full days between admission and discharge from the hospital. A calendar day will be counted toward the total only if the duration of stay on that day is two hours or longer.
Renal function recovery at hospital discharge | From enrollment to hospital discharge or 90 days (whichever occurs first)
  Recovery will be defined as improvement in kidney function based on serum creatinine value at hospital discharge compared with baseline serum creatinine.
  Baseline serum creatinine will be defined as either of the following (in order of priority) 1) Average of 3 closest outpatient values 7-365 days before index hospitalization; 2) Lowest value in the inpatient setting 7-365 days before index hospitalization; 3) Lowest value in the first 30 days during index hospitalization (not during or within 48h after RRT discontinuation).
  Patients who have serum creatinine <0.3 mg/dL higher than baseline at hospital discharge will be considered to have recovered renal function.
Renal function recovery at follow-up | From enrollment to 90-days post-ICU admission follow-up
  Recovery will be defined as improvement in kidney function based of serum creatinine value at follow-up compared with baseline serum creatinine.
  Baseline serum creatinine will be defined as either of the following (in order to priority) 1) Average of 3 closest outpatient values 7-365 days before index hospitalization; 2) Lowest value in the inpatient setting 7-365 days before index hospitalization; 3) Lowest value in the first 30 days during index hospitalization (not during or within 48h after RRT discontinuation).
  Patients who have serum creatinine <0.3 mg/dl higher than baseline at follow-up will be considered to have recovered renal function.
RRT dependence at hospital discharge | From RRT initiation to hospital discharge or 90 days (whichever occurs first)
  Patients will be classified as RRT-dependent if they continue to require any form of RRT at discharge. Patients who no longer require RRT will be classified as RRT-independent.
RRT dependence at follow-up | From RRT initiation (day 0) to 90-days post-ICU admission follow-up
  Patients will be classified as RRT-dependent if they continue to require any form of RRT at follow-up assessment. Patients who no longer require RRT will be considered RRT-independent.
Anticoagulation-related complications associated with RRT | RRT initiation (day 0) to RRT day 6 or RRT termination (whichever occurs first)
  These include complications attributable to different types of anticoagulation (systemic unfractionated heparin, systemic low molecular weight heparin, regional citrate anticoagulation, other) used during RRT. Events include hemorrhage, heparin-induced thrombocytopenia (where relevant), citrate excess (where relevant), and citrate deficit (where relevant).
Infectious complications associated with RRT | RRT initiation (day 0) to RRT day 6 or RRT termination (whichever occurs first)
  These include infections associated with RRT. Events include catheter-related bloodstream infections, catheter insertion-site infections, and secondary peritonitis.
RRT-related procedural complications | RRT initiation (day 0) to RRT day 6 or RRT termination (whichever occurs first)
  Procedural or mechanical complications occurring during RRT will be identified from medical records and bedside documentation. These include catheter malfunction (e.g., kinking, disconnection, malposition, migration, catheter tip adherence to vessel wall), circuit interruptions, circuit replacements, RRT downtime (where relevant).

CONTACTS AND LOCATIONS:
Overall Officials: Javier A Neyra, MD, MSCS, Principal Investigator — University of Alabama at Birmingham
Locations (13):
- Hospital Obrero No 2, Cochabamba, Bolivia
- Brazil (3):
  - Ana Nery Hospital, Bahia
  - Hospital Sao Lucas da PUCRS, Porto Alegre
  - Hospital das Clínicas da Universidade de São Paulo, São Paulo
- Hospital Las Higueras, Talcahuano, Chile
- Colombia (2):
  - Fundación Cardioinfantil, Bogotá
  - Hospital San Jose de Popayan, Popayán
- DIALNEF, Quito, Ecuador
- Instituto Guatemalteco de Seguridad Social, Guatemala City, Guatemala
- Mexico (3):
  - Hospital Civil de Guadalajara, Guadalajara
  - Hospital General de México Dr Eduardo Liceaga, Mexico City
  - Hospital Universitario "José Eleuterio González", Monterrey
- Hospital Nacional Arzobispo Loayza, Lima, Peru

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lombardi R, Rosa-Diez G, Ferreiro A, Greloni G, Yu L, Younes-Ibrahim M, Burdmann EA; Acute Kidney Injury Committee of the Latin American Society of Nephrology and Hypertension Working Group. Acute kidney injury in Latin America: a view on renal replacement therapy resources. Nephrol Dial Transplant. 2014 Jul;29(7):1369-76. doi: 10.1093/ndt/gfu078. Epub 2014 Apr 16. PMID 24744281
- [Background] Bello AK, McIsaac M, Okpechi IG, Johnson DW, Jha V, Harris DCH, Saad S, Zaidi D, Osman MA, Ye F, Lunney M, Jindal K, Klarenbach S, Kalantar-Zadeh K, Kovesdy CP, Parekh RS, Prasad B, Khan M, Riaz P, Tonelli M, Wolf M, Levin A; ISN North America and the Caribbean Regional Board. International Society of Nephrology Global Kidney Health Atlas: structures, organization, and services for the management of kidney failure in North America and the Caribbean. Kidney Int Suppl (2011). 2021 May;11(2):e66-e76. doi: 10.1016/j.kisu.2021.01.001. Epub 2021 Apr 12. PMID 33981472
- [Background] Wainstein M, Nlandu Y, Viecelli A, Neyra JA, Arruebo S, Caskey FJ, Damster S, Donner JA, Jha V, Levin A, Nangaku M, Saad S, Tonelli M, Ye F, Okpechi IG, Bello AK, Johnson DW, Cerda J. A global snapshot on health systems capacity for detection, monitoring, and management of acute kidney injury: A multinational study from the ISN-GKHA. PLOS Glob Public Health. 2024 Oct 15;4(10):e0003823. doi: 10.1371/journal.pgph.0003823. eCollection 2024. PMID 39405323
- [Background] Mehta RL, Burdmann EA, Cerda J, Feehally J, Finkelstein F, Garcia-Garcia G, Godin M, Jha V, Lameire NH, Levin NW, Lewington A, Lombardi R, Macedo E, Rocco M, Aronoff-Spencer E, Tonelli M, Zhang J, Remuzzi G. Recognition and management of acute kidney injury in the International Society of Nephrology 0by25 Global Snapshot: a multinational cross-sectional study. Lancet. 2016 May 14;387(10032):2017-25. doi: 10.1016/S0140-6736(16)30240-9. Epub 2016 Apr 13. PMID 27086173
- [Background] Rehman AU, Renzi S, Castro DAB, Cervantes L, Clavero R, Davidson B, Farias MR, Girard VC, Claure-Del Granado R, Ramirez-Guerrero G, Jimenez D, Leon Rabanal CP, Molano Trivino A, Reis T, Rizo-Topete L, Vega-Vega O, Viecelli AK, Kamile Singer Wallbach-Massai K, Wainstein M, Karam S, Neyra JA. Barriers and Facilitators to Renal Replacement Therapy for Acute Kidney Injury in Latin America: Insights From an Expert Roundtable. Kidney Int Rep. 2025 Jun 19;10(8):2515-2519. doi: 10.1016/j.ekir.2025.06.030. eCollection 2025 Aug. No abstract available. PMID 40814609
- [Background] Ponce D, Balbi A. Acute kidney injury: risk factors and management challenges in developing countries. Int J Nephrol Renovasc Dis. 2016 Aug 22;9:193-200. doi: 10.2147/IJNRD.S104209. eCollection 2016. PMID 27578995
- [Background] Susantitaphong P, Cruz DN, Cerda J, Abulfaraj M, Alqahtani F, Koulouridis I, Jaber BL; Acute Kidney Injury Advisory Group of the American Society of Nephrology. World incidence of AKI: a meta-analysis. Clin J Am Soc Nephrol. 2013 Sep;8(9):1482-93. doi: 10.2215/CJN.00710113. Epub 2013 Jun 6. PMID 23744003